CLINICAL TRIAL: NCT04315311
Title: A Phase 4 Open-Label Single-Arm Study To Evaluate The Use Of CREON In Subjects With EPI Due To Etiologies Other Than Cystic Fibrosis, Chronic Pancreatitis, Pancreatectomy, Or Pancreatic Cancer
Brief Title: Study Of Effects Of Oral CREON Capsules In Adult Participants With Exocrine Pancreatic Insufficiency Not Due To Cystic Fibrosis, Chronic Pancreatitis, Pancreatectomy, Or Pancreatic Cancer
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-112
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Exocrine Pancreatic Insufficiency (EPI)
Keywords: EPI; Exocrine pancreatic insufficiency; ABT-SLV245; Creon; Pancrelipase
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CREON (Experimental): Participants will receive daily dose of CREON.
  Interventions: Drug: CREON

INTERVENTIONS:
Drug: CREON — Capsule: Oral
  Other Names: Pancrelipase; ABT-SLV245

SUMMARY:
Exocrine pancreatic insufficiency (EPI) is a condition where the pancreas does not have enough pancreatic enzymes to break down food. Some symptoms of EPI are frequent gas/bloating, unexplained stomach pains, frequent diarrhea, and foul-smelling, greasy stools. The purpose of this study is to see how effective CREON is for treating symptoms of EPI due to causes other than cystic fibrosis (CF), chronic pancreatitis (CP), pancreatectomy (PY), or pancreatic cancer (PC).

CREON (Pancrelipase) is an approved drug used to treat people who cannot digest food normally due to their pancreas not making enough enzymes. Adult participants with a diagnosis of EPI due to causes other than CF, CP, PY, or PC will be enrolled. Around 50 participants will be enrolled in approximately 20 sites in the United States.

Participants will receive oral CREON capsules with each meal and snack beginning at Day 1 for 27 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or a clinic. Participants will need to be confined for 2 separate periods of 6 to 8 days each to measure Co-efficient of Fat Absorption (during screening and after enrollment). The effect of the treatment will be checked by medical assessments, blood and stool tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of exocrine pancreatic insufficiency (EPI).
* Participants who are on pancreatic enzyme replacement therapy (PERT) at the time of consent must have a clinical diagnosis of EPI by their physician.

Exclusion Criteria:

* History of cystic fibrosis, chronic pancreatitis, pancreatectomy, pancreatic cancer, or fibrosing colonopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-06 (Estimated); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Change In Coefficient Of Fat Absorption (CFA) From Baseline | Week 1
  CFA is calculated as 100*[fat intake - stool fat]/fat intake. Fat intake will be determined from fat content of food consumed on Days 3 to 5 in the confinement period. Stool fat will be determined from the fat content in the stool(s) collected between the two dye markers in the confinement period.

SECONDARY OUTCOMES:
Change In Gastrointestinal (GI) Symptoms From Baseline | Week 1
  Change in GI symptoms is measured by AbbVie exocrine pancreatic insufficiency (EPI) symptom questionnaire. EPI symptom questionnaire is a 12-item patient-reported outcome (PRO) instrument that assesses EPI symptoms over the past 7 days.
Change In Stool Frequency From Baseline | Week 1
  Stool frequency per 24 hours will be recorded daily during the 2 confinement periods. The average stool frequency per 24 hours during confinement period 1 will be considered as baseline.
Change In Stool Consistency From Baseline | Week 1
  Stool consistency will be evaluated using the Bristol Stool Scale. The Bristol Stool chart is a medical aid designed to classify feces.
Change In Vitamin D From Baseline | Up To Week 27
  Change from Baseline in vitamin D will be assessed through clinical laboratory testing.
Change In Vitamin E From Baseline | Up To Week 27
  Change from Baseline in vitamin E will be assessed through clinical laboratory testing.
Change In Vitamin K From Baseline | Up To Week 27
  Change from Baseline in vitamin K will be assessed through clinical laboratory testing.
Change In Vitamin A From Baseline | Up To Week 27
  Change from Baseline in vitamin A will be assessed through clinical laboratory testing.
Change In Retinol-Binding Protein From Baseline | Up To Week 27
  Change from Baseline in retinol-binding protein will be assessed through clinical laboratory testing.
Change In Albumin From Baseline | Up To Week 27
  Change from Baseline in albumin will be assessed through clinical laboratory testing.
Change In Prealbumin From Baseline | Up To Week 27
  Change from Baseline in prealbumin will be assessed through clinical laboratory testing.
Change In Transferrin From Baseline | Up To Week 27
  Change from Baseline in transferrin will be assessed through clinical laboratory testing.
Change In Weight From Baseline | Up To Week 27
  The mean change of weight from Baseline will be calculated.
Change In Body Mass Index (BMI) From Baseline | Up To Week 27
  BMI is a measure of body fat based on weight in relation to height.
Change In Hip Circumference From Baseline | Up To Week 27
  Hip circumference is measured by placing the measuring tape around the maximum circumference of the buttocks.
Change In Waist Circumference From Baseline | Up To Week 27
  Waist circumference is measured by placing a measuring tape on top of the hip bone and wrapping the tape around the waist.
Change In Gastrointestinal Quality Of Life Index (GIQLI) From Baseline | Up To Week 27
  GIQLI is a 36-item patient reported outcome (PRO) instrument used to assess GI-specific quality of life in participants with GI disorders, with response score ranging from 0 to 4 (0 being "all the time" and 4 being "never").

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: Related info — https://www.rxabbvie.com